CLINICAL TRIAL: NCT00829257
Title: A Proof of Concept Study to Evaluate the Additive Effects of HFA-BDP (Qvar) to Fluticasone/Salmeterol (Seretide) on Surrogate Markers of Small and Large Airway Inflammation in Refractory Asthma
Brief Title: Additive Effects of QVAR to (Seretide) on Surrogate Markers of Airway Inflammation in Refractory Asthma
Acronym: PAW01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PAW01; Eudract no: 2008-001811-40 (Registry Identifier: 2008RC10)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fine particle steroid inhaler (Experimental): HFA-BDP plus Fluticasone/Salmeterol Combination
  Interventions: Drug: HFA-BDP; Drug: Seretide
- Coarse Particle Inhaler (Active Comparator): FP plus Fluticasone/Salmeterol combination
  Interventions: Drug: Fluticasone; Drug: Seretide

INTERVENTIONS:
Drug: HFA-BDP — HFA-BDP (Qvar) 100ug 2puff b.i.d
  Arms: Fine particle steroid inhaler
Drug: Fluticasone — Fluticasone propionate Accuhaler 250ug b.i.d.
  Arms: Coarse Particle Inhaler
Drug: Seretide — Fluticasone/Salmeterol (Seretide) 500/50ug, 1 puff b.i.d

SUMMARY:
The purpose of this study is to establish whether addition of extra-fine particle steroid inhalers achieve additional suppression of small airways inflammation when added to 'standard' Fluticasone/Salmeterol combination therapy in refractory asthma.

ELIGIBILITY:
Inclusion Criteria:

* Refractory, non-smoking asthmatics with FEV1 les than 80% predicted
* RV greater than 100% predicted and CANO greater than 3ppb when stepped up to 1000µg of fluticasone per day, with or without additional asthma medication.
* Informed consent and ability to perform exhaled nitric oxide assessment.
* Participants must be on greater than 500mcg of fluticasone per day to enter dose ramp run-in.

Exclusion Criteria:

* Recent respiratory infection or oral steroid use.
* Pregnancy or lactation.
* Known or suspected contra-indication to any of the IMP's.
* CANO less than 3ppb, FEV1 greater than 80% or RV less than 100% at post-optimisation visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Alveolar nitric oxide | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Williamson, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, Ninewells Hospital and Medical School, Dundee, Scotland, United Kingdom

REFERENCES:
- [Result] Williamson PA, Short PM, Vaidyanathan S, Lipworth BJ. Inhaled and systemic corticosteroid response in severe asthma assessed by alveolar nitric oxide: a randomized crossover pilot study of add-on therapy. Br J Clin Pharmacol. 2013 Jan;75(1):93-102. doi: 10.1111/j.1365-2125.2012.04319.x. PMID 22568828